CLINICAL TRIAL: NCT05374473
Title: An Online Lifestyle Modification Course for People With MS: a Randomised Controlled Trial of Course Effectiveness
Brief Title: An Online Lifestyle Modification Course for People With Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Melbourne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 23458
Record Dates: First submitted 2022-04-25; First posted 2022-05-16 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Multiple Sclerosis
Keywords: Randomised controlled trial; Lifestyle modification; Online intervention
MeSH Terms: conditions — Multiple Sclerosis | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Two forms of the course were developed:
  1. an intervention course based delivering evidence based information regarding modifiable lifestyle related risk factors implicated in disease progression; and
  2. a standard-care course, similar in format and presentation, but containing general information sourced from standard MS websites.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention-tailored program with information regarding modifiable lifestyle related risk factors implicated in disease progression.
  Interventions: Behavioral: Lifestyle modification
- Standard-care (Other): containing general health information sourced from standard MS websites.
  Interventions: Behavioral: Standard-care

INTERVENTIONS:
Behavioral: Lifestyle modification — Content in the intervention arm was adapted from an evidence-based lifestyle modification program for people with MS outlined in print previously presented in a face-to-face format. The integrated lifestyle modification program translates the research evidence regarding modification of lifestyle related risk factors and health outcomes based on a detailed review of the literature around modifiable lifestyle risk factors that may influence MS disease progression, as outlined in the book Overcoming Multiple Sclerosis: the 7-step recovery program.
  Arms: Intervention
Behavioral: Standard-care — Content in standard-care arm was adapted from MS-related websites
  Arms: Standard-care

SUMMARY:
Lifestyle factors are known to affect the progression of multiple sclerosis (MS). Studies of participants with MS attending an evidence-based lifestyle modification program, delivered via face-to-face workshops, have demonstrated improved mental and physical health, reduced relapse rate and improved quality of life over 3 years follow up, and that behaviour change was feasible and sustainable. However, the face-to-face modality of this educational intervention is resource intensive, and accessibility may be impeded by geography, cost, and MS-specific factors such as illness, fatigue, and disability. Furthermore, the COVID-19 pandemic has highlighted the unpredictable ability to travel and the importance of flexibility of health-related education.

The Neuroepidemiology Unit at the University of Melbourne has developed the Multiple Sclerosis Online Course (MSOC) to deliver a widely accessible and user-friendly educational tool for people with MS. The course aims to deliver the best available evidence regarding lifestyle-related risk factors in the development and progression of MS and behaviour modification to improve health outcomes.

Two forms of the course were developed:

1. an intervention course delivering evidence-based information regarding modifiable lifestyle related risk factors implicated in disease progression; and
2. a standard-care course, similar in format and presentation, but containing general information sourced from standard MS websites. Both courses have seven modules delivered over six weeks.

A feasibility study involving the delivery of the intervention and standard-care course was conducted from April to June 2021. The study assessed the primary outcomes of attrition in both intervention and standard-care arm. Secondary outcomes assessed assessed learnability, accessibility, and desirability via a Likert scale follow-up survey. A qualitative analysis examining motivation, expectations and outcomes was also conducted. Tertiary outcomes assessed the completion of the baseline surveys, a requirement to enter the course. Based on the feasibility study, the investigators have modified recruitment strategies, functionality, and the community forum aspects of the course. Investigators now aim to test the effectiveness of the intervention arm of the course versus the standard-care arm in a larger randomised controlled trial.

Objective:

To prospectively examine whether an MS Online intervention course (intervention arm) can deliver an evidence-based educational intervention that results in behaviour change which can be sustained and translated into improved health outcomes for people with MS, and whether these effects are superior to the MS Online standard-care course (control arm).

Participants who are 18 or older, diagnosed with multiple sclerosis by a doctor are welcome to join our study.

The online course will run for 6 weeks. During this time, there are no formal assessments or minimum time investment required, which means participants are free to navigate the course as they see fit.

Prior to commencing the study, participants will be asked fill-out a survey about their health (e.g., fatigue) and lifestyle (e.g., diet) and will be asked to fill this out again during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to read, write, and speak English;
2. Be 18 years old or over;
3. Have a confirmed diagnosis of relapsing-remitting MS by a neurologist;
4. Be able to access the internet and be able to view sessions.

Exclusion Criteria:

1. Experiencing any serious co-morbid chronic illness or neurological illness/injury other than MS that would threaten regular participation or significantly affect the outcome measures in its own right, such as motor neurone disease or stroke, as determined by the study investigators;
2. Currently participating in another study or self-management program involving modification of lifestyle.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 945 (Actual)
Dates: Start 2022-06-24 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in physical health-related quality of life from baseline to 6- 12- and 30-month follow-up | Pre-intervention (Baseline) to post-intervention (6-, 12- and 30-month follow-up)
  Health-related quality of life will be measured using the Multiple Sclerosis Quality of Life survey (MSQOL-54) (Vickrey, Hays, Harooni, Myers, & Ellison, 1995). The MSQoL-54 is a psychometrically validated, MS-specific, multi-dimensional inventory of patient-centered health status, and consists of 54 questions on items relevant to people with Multiple Sclerosis in the areas of health distress, sexual function, satisfaction with sexual function, overall quality of life, cognitive function, energy, and pain and social function. A physical and a mental dimension underlie the MSQOL-54: the Physical Health Composite (PHC) and Mental Health Composite (MHC). PHC scores range from 0 to 100, where higher values indicate better physical quality of life. Changes in PHC scores (from baseline to 6- 12- and 30-month follow-up) will be assessed and compared between participants in the intervention and standard care groups.
Change in mental health-related quality of life from baseline to 6- 12- and 30-month follow-up | Pre-intervention (Baseline) to post-intervention (6-, 12- and 30-month follow-up)
  Health-related quality of life will be measured using the Multiple Sclerosis Quality of Life survey (MSQOL-54)(Vickrey, Hays, Harooni, Myers, & Ellison, 1995). The MSQoL-54 is a psychometrically validated, MS-specific, multi-dimensional inventory of patient-centered health status, and consists of 54 questions on items relevant to people with Multiple Sclerosis in the areas of health distress, sexual function, satisfaction with sexual function, overall quality of life, cognitive function, energy, and pain and social function. A physical and a mental dimension underlie the MSQOL-54: the Physical Health Composite (PHC) and Mental Health Composite (MHC). MHC scores range from 0 to 100, where higher values indicate better mental quality of life. Changes in MHC scores (from baseline to 6- 12- and 30-month follow-up) will be assessed and compared between participants in the intervention and standard care groups.

SECONDARY OUTCOMES:
Change in depression | Pre-intervention (Baseline) to post-intervention (6-, 12- and 30-month follow-up)
  Participants in the intervention group will be compared to those in the standard-care group on their changes in depression from baseline to 6-, 12- and 30-month follow-up. The Hospital Anxiety and Depression Scale (HADS) is used to measure depressive symptoms. The HADS is commonly used for screening for anxiety and depression, as well as selecting and monitoring treatment and has been used to measure anxiety and depression in Multiple Sclerosis (Zigmond & Snaith, 1983). The HADS contains 14 items and consists of two subscales: anxiety and depression. The depression subscale ranges from 0 to 21 points. Scores of 11 or more indicate a significant condition of depression, with scores of 8-10 represents 'mild to moderate' and 0-7 'no depression'. Changes in depression (increased or decreased depression scores and shifted depression classification) will be assessed and compared between participants in the intervention and standard care groups.
Change in anxiety | Pre-intervention (Baseline) to post-intervention (6-, 12- and 30-month follow-up)
  Participants in the intervention group will be compared to those in the standard-care group on their changes in anxiety, from baseline to 6-, 12- and 30-month follow-up. The Hospital Anxiety and Depression Scale (HADS) is used to measure anxiety. The HADS is commonly used for screening for anxiety and depression, as well as selecting and monitoring treatment and has been used to measure anxiety and depression in Multiple Sclerosis (Zigmond & Snaith, 1983). The HADS contains 14 items and consists of two subscales: anxiety and depression. The anxiety subscale ranges from 0 to 21 points. Scores of 11 or more indicate a significant condition of anxiety, with scores of 8-10 represents 'mild to moderate' and 0-7 'no anxiety'. Changes in anxiety (increased or decreased anxiety scores or shifted anxiety classification) will be assessed and compared between participants in the intervention and standard care groups.
Change in fatigue | Pre-intervention (Baseline) to post-intervention (6-, 12- and 30-month follow-up)
  Participants in the intervention group will be compared to those in the standard-care group on changes in fatigue from baseline to 6-, 12- and 30-month follow-up. Fatigue will be measured by the 9-item Fatigue Severity Scale (FSS)(Krupp, LaRocca, Muir-Nash, & Steinberg, 1989). The FSS has mean score range from 1-7, with higher score indicates more fatigue. A mean score ≥ 4 will be used as a cut-off to indicate clinically significant fatigue. A meaningful change on the FSS has been reported demonstrated to be a change of ≥1.9 points in people with MS (Learmonth et al., 2013) and so here a change in mean score of 1.9 points or more will be considered clinically meaningful. Changes in fatigue (increased or decreased fatigue scores or shifted fatigue classification) will be assessed and compared between participants in the intervention and standard care groups.
Change in disability | Pre-intervention (Baseline) to post-intervention (6-, 12- and 30-month follow-up)
  Participants in the intervention group will be compared to those in the standard-care group on their changes in level of disability, from baseline to 6-, 12- and 30-month follow-up. The Patient-Determined Disease Steps (PDDS) will be used to measure disability (Hohol, Orav, &Weiner, 1999). The PDDS is a self-reported measure of disability, scored ordinally from 0 (normal) to 8 (bed bound) with detail descriptors and definitions. Changes in disability (increased or decreased PDDS scores) will be assessed and compared between participants in the intervention and standard care groups.
Change in self-efficacy | Pre-intervention (Baseline) to post-intervention (6-, 12- and 30-month follow-up)
  Participants in the intervention group will be compared to those in the standard-care group on changes in self-efficacy (the belief in one's ability to produce the effects or outcomes one wants). Self-efficacy will be measured using the University of Washington Self-Efficacy (UWSE) survey, a psychometrically sound instrument that includes 6 items for measuring self-efficacy, validated in MS (Amtmann et al., 2012). UWSE MS total score range from 6 to 30, higher scores indicate higher self-efficacy. Total scores will be converted to standardised T-scores, which have a mean of 50 and standard deviation of 10. Higher T-scores indicate greater self-efficacy. Changes in self-efficacy (increased or decreased T-scores) will be assessed and compared between participants in the intervention and standard care groups.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra L Neate, Doctor, Principal Investigator — University of Melbourne
Locations (1):
- The University of Melbourne, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jelinek, G. (2016). Overcoming multiple sclerosis: the evidence-based 7 step recovery program. Atlantic Books.
- [Background] Marck CH, De Livera AM, Brown CR, Neate SL, Taylor KL, Weiland TJ, Hadgkiss EJ, Jelinek GA. Health outcomes and adherence to a healthy lifestyle after a multimodal intervention in people with multiple sclerosis: Three year follow-up. PLoS One. 2018 May 23;13(5):e0197759. doi: 10.1371/journal.pone.0197759. eCollection 2018. PMID 29791509
- [Result] Hadgkiss EJ, Jelinek GA, Weiland TJ, Pereira NG, Marck CH, van der Meer DM. The association of diet with quality of life, disability, and relapse rate in an international sample of people with multiple sclerosis. Nutr Neurosci. 2015 Apr;18(3):125-36. doi: 10.1179/1476830514Y.0000000117. Epub 2014 Mar 17. PMID 24628020
- [Result] Vickrey BG, Hays RD, Harooni R, Myers LW, Ellison GW. A health-related quality of life measure for multiple sclerosis. Qual Life Res. 1995 Jun;4(3):187-206. doi: 10.1007/BF02260859. PMID 7613530
- [Result] Krupp LB, LaRocca NG, Muir-Nash J, Steinberg AD. The fatigue severity scale. Application to patients with multiple sclerosis and systemic lupus erythematosus. Arch Neurol. 1989 Oct;46(10):1121-3. doi: 10.1001/archneur.1989.00520460115022. PMID 2803071
- [Result] Learmonth YC, Dlugonski DD, Pilutti LA, Sandroff BM, Motl RW. The reliability, precision and clinically meaningful change of walking assessments in multiple sclerosis. Mult Scler. 2013 Nov;19(13):1784-91. doi: 10.1177/1352458513483890. Epub 2013 Apr 15. PMID 23587605
- [Result] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Result] Hohol MJ, Orav EJ, Weiner HL. Disease steps in multiple sclerosis: a longitudinal study comparing disease steps and EDSS to evaluate disease progression. Mult Scler. 1999 Oct;5(5):349-54. doi: 10.1177/135245859900500508. PMID 10516779
- [Result] Amtmann D, Bamer AM, Cook KF, Askew RL, Noonan VK, Brockway JA. University of Washington self-efficacy scale: a new self-efficacy scale for people with disabilities. Arch Phys Med Rehabil. 2012 Oct;93(10):1757-65. doi: 10.1016/j.apmr.2012.05.001. Epub 2012 May 7. PMID 22575393

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-13): https://cdn.clinicaltrials.gov/large-docs/73/NCT05374473/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT05374473/ICF_001.pdf